CLINICAL TRIAL: NCT01637636
Title: An Open-label, Single-sequence Study in Two Cohorts of Healthy Subjects to Evaluate the Single-dose Pharmacokinetics of Tasimelteon Alone and in Combination With a CYP3A4 Inhibitor, Ketoconazole, or a CYP3A4 Inducer, Rifampin.
Brief Title: Pharmacokinetics of Tasimelteon Alone and in Combination With a CYP3A4 Inhibitor, Ketoconazole, or a CYP3A4 Inducer, Rifampin.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1112
Record Dates: First submitted 2012-06-28; First posted 2012-07-11 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: rifampin,; ketoconazole,; CYP3A4,; tasimelteon,; VEC-162; Pharmacokinetics
MeSH Terms: interventions — tasimelteon; Rifampin; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifampin (Experimental)
  Interventions: Drug: tasimelteon; Drug: Rifampin
- Ketoconazole (Experimental)
  Interventions: Drug: tasimelteon; Drug: Ketoconazole

INTERVENTIONS:
Drug: tasimelteon — 20mg, oral capsule, once, Days 1 and 12
  Other Names: VEC-162, BMS-214778
  Arms: Rifampin
Drug: tasimelteon — 20mg, oral capsule, once, Days 1 and 6
  Other Names: VEC-162, BMS-214778
  Arms: Ketoconazole
Drug: Rifampin — 600mg, oral capsules (2 x 300mg), once daily (QD), Days 2-11
  Arms: Rifampin
Drug: Ketoconazole — 400mg, oral tablets (2 x 200mg), once daily (QD), Days 2-6
  Arms: Ketoconazole

SUMMARY:
The purpose of this research study is to understand whether there is any difference in the amount of tasimelteon (including its breakdown product) in the blood when taken alone and in combination with either rifampin or ketoconazole.

Cytochrome P450 3A4 is an important enzyme produced by the body to breakdown certain medications. In this study, the effect that this important enzyme has on tasimelteon is being studied by assessing the effect rifampin and ketoconazole have on tasimelteon and how they are broken down by your body. Rifampin is a known inducer of Cytochrome P450 3A4 enzyme meaning that it increases the activity of the enzyme. Ketoconazole is a known inhibitor of Cytochrome P450 3A4 enzyme meaning that it decreases the activity of the enzyme.

In addition, the safety and tolerability of tasimelteon will also be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18 - 55 years, inclusive;
2. Non-smokers;
3. Subjects with Body Mass Index (BMI) of ≥18 and ≤35 kg/m^2;
4. Males, non-fecund females, or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing;
5. Vital signs which are within the ranges shown below:

   1. Body temperature between 35.0-37.5 °C;
   2. Systolic blood pressure between 90-150 mmHg;
   3. Diastolic blood pressure between 50-95 mmHg;
   4. Pulse rate between 50-100 bpm.
6. Ability and acceptance to provide written informed consent;
7. Willing and able to comply with study requirements and restrictions;
8. In good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests and urinalysis;

Exclusion Criteria:

1. History of recent (within six months) drug or alcohol abuse;
2. Any major surgery within three months of Baseline or any minor surgery within one month;
3. History or current evidence of cardiovascular, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction or psychiatric disease judged by the Investigator to be clinically significant;
4. History (including family history) or current evidence of congenital long QT syndrome or known acquired QT interval prolongation;
5. Subjects who are currently considered a suicide risk, any subject who has ever made a suicide attempt, or those who are currently demonstrating active (within the past 6 months) suicidal ideation;
6. Any condition requiring the regular use of medication except those listed in Section 8.2 of the protocol;
7. Exposure to any investigational drug, including placebo, within 30 days or 5 half-lives (whichever is longer) of baseline
8. Exposure (within 2 weeks of the Baseline Visit) to any over-the-counter medications including melatonin, dietary supplements and/or herbal remedies, except those listed on Section 8.2;
9. Treatment with any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 days preceding the Screening visit;
10. History of intolerance and/or hypersensitivity to ketaconazole, drugs similar to ketoconazole (e.g. miconzaole or fluconazole), rifampin, tasimelteon, and/or drugs similar to tasimelteon including melatonin;
11. Donation or loss of 400 mL or more of blood within one month prior to the Baseline Visit;
12. Significant illness within the two weeks prior to Baseline;
13. Pregnant or lactating females;
14. History of porphyria or liver disease and/or positive for one or more of the following serological results:

    1. A positive hepatitis C antibody test (anti-HCV)
    2. A positive hepatitis B surface antigen (HBsAg)
    3. A positive HIV test result
15. Participation in a previous BMS-214778/VEC-162 trial;
16. Use of any food or beverage containing grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g. kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens) and charbroiled meats for at least 2 weeks before the Baseline Visit until the end of the study;
17. Inability to be venipunctured and/or tolerate venous access;
18. Subjects who are unable to read or speak English;
19. Any other sound medical reason as determined by the clinical Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of tasimelteon and tasimelteon's metabolites with and without the CYP3A4 inhibitor ketoconazole. | Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose. Days 6 and 7: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of tasimelteon and tasimelteon's metabolites with and without the CYP3A4 inducer rifampin. | Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose. Days 12 and 13: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Bio-Kinetic Clinical Applications, Springfield, Missouri, United States